CLINICAL TRIAL: NCT05769244
Title: Near Infrared Spectroscopy and Testicular Torsion in Children
Acronym: SPIRETTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PI2019_843_0053
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Diagnostic Test; NIRS; Testicular Torsion; Diagnosis; Child
MeSH Terms: conditions — Spermatic Cord Torsion; Disease | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- testicular torsion (Experimental)
  Interventions: Other: near-infrared spectroscopy (NIRS)
- other testicular pathology (Active Comparator)
  Interventions: Other: near-infrared spectroscopy (NIRS)
- healthy patients (Sham Comparator)
  Interventions: Other: near-infrared spectroscopy (NIRS)

INTERVENTIONS:
Other: near-infrared spectroscopy (NIRS) — NIRS measurements will be performed on each testicle on a group of healthy boys and on a group of boys under 18 years consulting to emergency for scrotal pain

SUMMARY:
NIRS estimates tissue saturation of oxygenation in tissue beds. Animals studies suggested that transscrotal NIRS measurements can quantify testicular hypoxia and differentiate between torsed and non torsed testicles. The results of human studies are not conclusive. The hypothesis is that the difference in NIRS values between torsed and healthy testicles would not be zero and that this difference would be zero in control group and that NIRS could help to detect rapidly a TT Testicular torsion (TT) is a functional emergency. The diagnosis is sometimes difficult to make. No paraclinical examination can eliminate it with certainty. The investigators aimed to evaluate the interest of transscrotal near-infrared spectroscopy (NIRS) for the diagnosis of TT of child

ELIGIBILITY:
Inclusion Criteria:

* Step 1: healthy boys between 0 and 16 years old
* Step 2Testicular pain group (Group 1 and 2): boy under 18 years, testicular pain

Exclusion Criteria:

* cutaneous scrotal lesion,
* fever (for the control group),
* hypertension

Max Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — NIRS measurement on testicules
Enrollment: 55 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
mean tissue oxygenation percentage (NIRS measurements) of the testicles for healthy boys | one day
  Near-infrared spectroscopy (NIRS) is a noninvasive technology that continuously monitors regional tissue oxygenation. Originally used for assessment of oxygen saturation of the brain, its use has now been expanded to evaluation of oxygenation of tissues other than the brain.
  Normal values for NIRS values are between 60-75% but physiological values of 55-60% have been reported in some cardiac patients
mean tissue oxygenation percentage (NIRS measurements) of the both testicles for boys with scrotal pain | one day
  Near-infrared spectroscopy (NIRS) is a noninvasive technology that continuously monitors regional tissue oxygenation. Originally used for assessment of oxygen saturation of the brain, its use has now been expanded to evaluation of oxygenation of tissues other than the brain.
  Normal values for NIRS values are between 60-75% but physiological values of 55-60% have been reported in some cardiac patients
mean tissue oxygenation percentage (NIRS measurements) between both testicles for boys with scrotal pain | one day
  Near-infrared spectroscopy (NIRS) is a noninvasive technology that continuously monitors regional tissue oxygenation. Originally used for assessment of oxygen saturation of the brain, its use has now been expanded to evaluation of oxygenation of tissues other than the brain.
  Normal values for NIRS values are between 60-75% but physiological values of 55-60% have been reported in some cardiac patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No